CLINICAL TRIAL: NCT06745271
Title: A Phase I, Open-label Study to Evaluate the Absorption, Metabolism, and Excretion and to Assess the Absolute Bioavailability Following a Single Oral Dose of [14C]-Tebapivat and Concomitant Single Intravenous Microdose of [13C2,15N3]-Tebapivat to Healthy Male Participants
Brief Title: A Study to Determine How Tebapivat is Absorbed, Broken Down, and Removed From the Body and the Extent to Which Tebapivat is Made Available in the Body in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG946-C-004
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-tebapivat and [13C2,15N3]-tebapivat (Experimental): Participants will receive a single oral dose of 10 milligrams (mg) [14C]-tebapivat containing 200 microcurie [μCi] of radiocarbon in a capsule followed by a single intravenous (IV) microdose of 0.1 mg [13C2,15N3]-tebapivat on Day 1.
  Interventions: Drug: [14C]-tebapivat; Drug: [13C2,15N3]-tebapivat

INTERVENTIONS:
Drug: [14C]-tebapivat — Oral Capsule
Drug: [13C2,15N3]-tebapivat — Intravenous Solution

SUMMARY:
The primary purpose of this study is to determine the routes, rates of elimination, mass balance of total radioactivity and metabolite profiles following a single oral dose of [14C]-tebapivat. To characterize the PK of tebapivat and [13C2,15N3]-tebapivat and determine the absolute bioavailability following single oral dose of [14C]-tebapivat relative to single intravenous microdose of [13C2,15N3]-tebapivat to healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male, of any race, between 18 and 55 years of age, inclusive.

   a. Males must agree to use contraception.
2. Body mass index between 18.0 and 30.0 kilograms per meter square (kg/m2), inclusive, and a body weight between 50 and 100 kilograms (kg), inclusive.
3. In good health, as determined by no clinically significant findings from medical history, 12-lead ECG and vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in, and from the physical examination at check-in, as assessed by the investigator or designee.
4. History of a minimum of 1 bowel movement per day.
5. Able to comprehend and are willing to sign the informed consent form (ICF) and abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, as determined by the investigator or designee.
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair are allowed; cholecystectomy is not allowed).
4. Positive hepatitis panel and/or positive human immunodeficiency virus test. Participants whose results are compatible with prior immunization may be included.
5. Administration of any vaccine within 30 days prior to dosing.
6. Use or intend to use any medications/products known to alter drug absorption, metabolism, and excretion (AME) processes, including St. John's wort, within 30 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
7. Use or intend to use any prescription medications/products within 14 days or 5 half-lives (whichever is longer) prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
8. Use or intend to use any slow release medications/products considered to still be active within 14 days or 5 half-lives (whichever is longer) prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
9. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to dosing, considered to potentially impact participant safety or the objectives of the study, as determined by the investigator or designee.
10. Participation in a clinical study involving administration of an IMP (new chemical entity) in the past 30 days or 5 half-lives of that drug (if known) prior to dosing, whichever is longer.
11. Have previously completed or withdrawn from this study or any other study investigating tebapivat and have previously received tebapivat.
12. Participants who have previously been dosed in >1 radiolabeled drug study in the last 12 months. For participants who have previously been dosed in 1 radiolabeled drug study within the last 12 months, the previous radiolabeled dose must be at least 6 months prior to check-in at the clinical research unit (CRU). The total 12 month exposure from this study and a maximum of 1 other previous radiolabeled study must be within the Code of Federal Regulations (CFR) recommended levels considered safe, per United States (US) Title 21 CFR 361.1.
13. Alcohol consumption of >21 units per week. One unit of alcohol equals 12 ounces (oz) (360 milliliters (mL)) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
14. Positive urine drug screen at screening or positive alcohol test result or positive urine drug screen at check-in.
15. History of alcoholism or drug/chemical abuse within 2 years prior to check-in.
16. Use of tobacco- or nicotine-containing products within 3 months prior to check-in, or positive cotinine at screening or check-in.
17. Receipt of blood products within 2 months prior to check-in.
18. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
19. Poor peripheral venous access.
20. Participants with exposure to significant diagnostic or therapeutic radiation (e.g., serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
21. Participants who, in the opinion of the investigator or designee, should not participate in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Radioactive Dose Excreted in Urine Over a Time Interval (feut1-t2) of [14C]-Tebapivat | Up to Day 42
Percentage of Radioactive Dose Excreted in Feces Over a Time Interval (fef t1-t2) of [14C]-Tebapivat | Up to Day 42
Cumulative Percentage of Radioactive Dose Excreted in Urine Over a Time Interval (Cum feut1-t2) of [14C]-Tebapivat | Up to Day 42
Cumulative Percentage of Radioactive Dose Excreted in Feces Over a Time Interval (Cum fef t1-t2) of [14C]-Tebapivat | Up to Day 42
Percentage of Total Radioactivity in Total Excreta (Feces + Urine) (Cum fe) of [14C]-Tebapivat | Up to Day 42
Amount of Drug Excreted in Urine (Aeu) of [14C]-Tebapivat | Up to Day 42
Cumulative Amount of Drug Excreted in Urine (Cum Aeu) of [14C]-Tebapivat | Up to Day 42
Renal Clearance (CLR) of [14C]-Tebapivat | Up to Day 42
Area Under the Concentration-Time Curve (AUC) From Time 0 to 168 Hours Postdose (AUC0-168) in Plasma for [14C]-Tebapivat and [13C2,15N3]-Tebapivat | Up to Day 7
AUC0-168 in Plasma and Whole Blood for Total Radioactivity | Up to Day 7
AUC From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-t) in Plasma for [14C]-Tebapivat and [13C2,15N3]-Tebapivat | Up to Day 21
AUC0-t in Plasma and Whole Blood for Total Radioactivity | Up to Day 42
AUC Extrapolated to Infinity (AUC0-inf) in Plasma for [14C]-Tebapivat and [13C2,15N3]-Tebapivat | Up to Day 21
(AUC0-inf) in Plasma and Whole Blood for Total Radioactivity | Up to Day 42
Maximum Observed Plasma Concentration (Cmax) for [14C]-Tebapivat and [13C2,15N3]-Tebapivat | Up to Day 21
Cmax in Plasma and Whole Blood for Total Radioactivity | Up to Day 42
Time to Reach Cmax (Tmax) for [14C]-Tebapivat and [13C2,15N3]-Tebapivat | Up to Day 21
Tmax in Plasma and Whole Blood for Total Radioactivity | Up to Day 42
Terminal Elimination Half-Life (t1/2) in Plasma for [14C]-Tebapivat and [13C2,15N3]-Tebapivat | Up to Day 21
T1/2 in Plasma and Whole Blood for Total Radioactivity | Up to Day 42
Ratio of AUC0-inf for Tebapivat to AUC0-inf for Total Radioactivity in Plasma | Up to Day 42
Ratio of AUC0-inf for Total Radioactivity in Whole Blood to AUC0-inf for Total Radioactivity in Plasma | Up to Day 42
Total Clearance Following IV Administration (CL) of [13C2,15N3]-Tebapivat | Up to Day 21
Apparent Volume of Distribution During the Terminal Phase Following IV Administration (Vz) of [13C2,15N3]-Tebapivat | Up to Day 21
Apparent Volume of Distribution at Steady State Following IV Administration (Vss) of [13C2,15N3]-Tebapivat | Up to Day 21
Ratio of Dose-Normalized AUC0-inf of Oral Administration of [14C]-Tebapivat Relative to IV Administration of [13C2,15N3]-Tebapivat | Up to Day 21
Quantitation of Major Metabolites of [14C]-Tebapivat in Plasma After Oral Administration | Up to Day 21
  Quantification of major metabolites of [14C]-tebapivat in plasma.
Quantitation of Major Metabolites of [14C]-Tebapivat in Excreta After Oral Administration | Up to Day 42
  Quantification of major metabolites of [14C]-tebapivat in excreta.
Identification of Chemical Structure of Major Metabolites of [14C]-Tebapivat in Plasma After Oral Administration | Up to Day 21
  Identification of the chemical structures of major metabolites of [14C]-tebapivat in plasma.
Identification of Chemical Structure of Major Metabolites of [14C]-Tebapivat in Excreta After Oral Administration | Up to Day 42
  Identification of the chemical structures of major metabolites of [14C]-tebapivat in excreta.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) by Type, Severity, and Relationship to Study Drug | Up to Day 28
Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Assessments | Baseline up to Day 28
Number of Participants With Clinically Significant Change From Baseline in Abnormal 12-Lead Electrocardiogram (ECG) Parameters | Baseline up to Day 28
Number of Participants With Clinically Significant Change From Baseline in Abnormal Vital Signs Measurements | Baseline up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Taha El-Shahat, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No